CLINICAL TRIAL: NCT05016362
Title: Patient Satisfaction After Medial Fat Pad Preservation in Upper Eyelid Blepharoplasty
Brief Title: Medial Fat Pad Preservation in Upper Eyelid Blepharoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Associate Professor, Benha University
Other Study IDs: Hamaky16
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Eyelid Diseases
Keywords: upper eyelid pad fat; blepharoplasty
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: blepharoplasty with repositioning of the nasal fat pad to the central arcus marginalis of the superior orbital rim during surgery.
  Interventions: Procedure: medial fat preservation upper blepharoplasty
- Group B: blepharoplasty with repositioning of the nasal fat pad to orbitoglabellar groove during surgery.
  Interventions: Procedure: medial fat preservation upper blepharoplasty

INTERVENTIONS:
Procedure: medial fat preservation upper blepharoplasty — medial fat preservation upper blepharoplasty increasing volumetric upper eyelid skin fold

SUMMARY:
Medial upper eyelid pad of fat bulge is a common problem. medial fat pad preservation might be a good adjutant to upper eyelid blepharoplasty

DETAILED DESCRIPTION:
Blepharoplasty with repositioning of the nasal fat pad to the central arcus marginalis of the superior orbital rim during surgery or orbitoglabellar groove

ELIGIBILITY:
Inclusion Criteria:

* upper eyelid medial pad of fat bulge

Exclusion Criteria:

* Other eyelid diseases and previous eyelid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: at least 18 years old participant with dermtochlasis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
global aesthetic improvement scale | 1 year
  calculate scale score (1-5);score 1:exceptional improvement and score 5 :worsened patient

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Elahamky, Principal Investigator — Benha university faculty of medicine
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates